CLINICAL TRIAL: NCT06532968
Title: Clinical Evaluation of Orion Lamina Cover in Patients Undergoing Lumbar Laminectomy With Instrumented Fusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orion Biotech Inc. (Industry)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-10-006C
Record Dates: First submitted 2024-07-30; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Degenerative Lumbar Spinal Stenosis; Degenerative Spondylolisthesis; Spinal Stenosis; Scoliosis; Spinal Fracture
MeSH Terms: conditions — Spinal Stenosis; Scoliosis; Spinal Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Sham Comparator): General spinal system
  Interventions: Device: Sham
- LMC group (Experimental): General spinal system with ORION spinal lamina cover
  Interventions: Device: ORION spinal lamina cover

INTERVENTIONS:
Device: Sham — Sham
  Arms: Control group
Device: ORION spinal lamina cover — an artificial lamina coverage of the ORION spinal system
  Arms: LMC group

SUMMARY:
Laminectomy with internal fixation and osseofusion is a common surgery for treating degenerative spinal diseases. It removes excessive bone spurs and removes the lamina for decompression to relieve nerve compression, and then utilizes a spinal fixation system to stabilize the structure to relieve lower limb pain, paralysis, and other symptoms. However, the spinal cord that lacks lamina coverage after surgery is often compressed by scar tissue formation and hematoma, leading to postoperative back and lower limb pain. Therefore, this trial is divided into two groups, comparing the use of the cross connector of the ORION spinal system - the spinal lamina cover and the general spinal fixation system (without lamina cover). For participants undergoing laminectomy with internal fixation and osseofusion, after utilizing the spinal lamina cover of the ORION spinal system, whether the nerve compression caused by postoperative scar tissue formation and hematoma can be effectively reduced, and the pain in the back and lower limbs can be improved.

ELIGIBILITY:
Inclusion Criteria:

* Gender and age: females and males are at least 20 years old
* Who with degenerative lumbar spondylolisthesis in one or two consecutive segments from lumbar vertebra L1 to sacral vertebra S1, and have objective evidence of back pain and numbness radiating to the lower limbs.
* Clinical symptoms of degenerative lumbar spondylolisthesis, accompanied by objective symptoms of neurological deficit; spinal stenosis, neurogenic claudication or bilateral radiating pain.
* Have received at least 3 months of non-surgical treatment without effectiveness.
* Radiographic examination was consistent with clinical symptoms of degenerative spondylolisthesis or spinal stenosis.
* After diagnosis who needs laminectomy with internal fixation and osseofusion
* Able and willing to sign the consent form and answer the questionnaire.

Exclusion Criteria:

* Already had lumbar surgery at the same lumbar vertebra
* Physically health not well
* Probably pregnant
* Who suffering from malignant tumors or infections
* below 20 years old
* Unable and unwilling to answer the questionnaire and return to the hospital for treatment
* Unable to undergo MRI examination due to any reason, such as having a cardiac rhythm regulator, ferromagnetic implants, or claustrophobia.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Magnetic Resonance Imaging (MRI) | Six months after surgery
  To observe the recovery of the participants' spine
Visual Analogue Scale (VAS) | Pre-surgery; one month after surgery; three months after surgery; six months after surgery
  To measure the pain and numb of the participants' back and limbs

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | Pre-surgery; one month after surgery; three months after surgery; six months after surgery
  To evaluate the functional disability of the participants' limbs
Sort Form-12 Health Survey (SF-12) | Pre-surgery; one month after surgery; three months after surgery; six months after surgery
  To evaluate the physical health of the participants

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Cheng Yao, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan